CLINICAL TRIAL: NCT03849287
Title: An Open-label, Randomized, Fasted, Single-dose, Three-way Crossover Study to Compare the Pharmacokinetic Characteristics and Safety Between Administration of CKD-333 and Coadministration of CKD-330 and D090 in Healthy Male Adults
Brief Title: Compare the Pharmacokinetics and Safety of CKD-333 With Co-administration CKD-330 and D090 in Healthy Male Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 170PK18039
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): * Period 1: CKD-333, formula I
  * Period 2: CKD-333, formula II
  * Period 3: CKD-330, D090
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090
- Group 2 (Experimental): * Period 1: CKD-333, formula I
  * Period 2: CKD-330, D090
  * Period 3: CKD-333, formula II
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090
- Group 3 (Experimental): * Period 1: CKD-333, formula II
  * Period 2: CKD-330, D090
  * Period 3: CKD-333, formula I
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090
- Group 4 (Experimental): * Period 1: CKD-333, formula II
  * Period 2: CKD-333, formula I
  * Period 3: CKD-330, D090
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090
- Group 5 (Experimental): * Period 1: CKD-330, D090
  * Period 2: CKD-333, formula I
  * Period 3: CKD-333, formula II
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090
- Group 6 (Experimental): * Period 1: CKD-330, D090
  * Period 2: CKD-333, formula II
  * Period 3: CKD-333, formula I
  Interventions: Drug: CKD-333, formula I; Drug: CKD-333, formula II; Drug: CKD-330, D090

INTERVENTIONS:
Drug: CKD-333, formula I — Test drug
Drug: CKD-333, formula II — Test drug
Drug: CKD-330, D090 — Reference Drug

SUMMARY:
The object of clinical trial is to investigate the pharmacokinetics and safety compared to CKD-333 and co-administration CKD-330, D090 under fasting condition in healthy male adults.

DETAILED DESCRIPTION:
An open-label, randomized, fasted, single-dose, three-way crossover study to compare the pharmacokinetic characteristics and safety between administration of CKD-333 and coadministration of CKD-330 and D090 in healthy male adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults aged 19 to 45 years
2. Body weight more than 50kg and within ideal body weight ±20%
3. signed informed consent form

Exclusion Criteria:

1. Have clinical significant medical history or disease that cardiovascular system, respiratory system, kidney, endocrine system, hematological system, digestive system , mental illness
2. Have a gastrointestinal disease history that can effect drug absorption or surgery
3. Systolic Blood pressure≥140mmHg or Systolic Blood pressure<90mmHg, Diastolic Blood Pressure≥90mmHg or Diastolic Blood Pressure<60mmHg

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2019-03-29 (Estimated); Study Completion 2019-04-06 (Estimated)

PRIMARY OUTCOMES:
AUClast of Candesartan | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Candesartan
AUClast of Amlodipine | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Amlodipine
AUClast of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Atorvastatin
Cmax of Candesartan | 0 hour ~ 72 hour after drug administration
  Maximum plasma concentration of Candesartan
Cmax of Amlodipine | 0 hour ~ 72 hour after drug administration
  Maximum plasma concentration of Amlodipine
Cmax of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Maximum plasma concentration of Atorvastatin

SECONDARY OUTCOMES:
AUCinf of Candesartan | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Candesartan
AUCinf of Amlodipine | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Amlodipine
AUCinf of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Atorvastatin
AUCinf of 2-hydroxy atorvastatin | 0 hour ~ 72 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of 2-hydroxy atorvastatin
Tmax of Candesartan | 0 hour ~ 72 hour after drug administration
  Time to maximum plasma concentration of Candesartan
Tmax of Amlodipine | 0 hour ~ 72 hour after drug administration
  Time to maximum plasma concentration of Amlodipine
Tmax of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Time to maximum plasma concentration of Atorvastatin
Tmax of 2-hydroxy atorvastatin | 0 hour ~ 72 hour after drug administration
  Time to maximum plasma concentration of 2-hydroxy atorvastatin
T1/2 of Candesartan | 0 hour ~ 72 hour after drug administration
  Half-life of Candesartan
T1/2 of Amlodipine | 0 hour ~ 72 hour after drug administration
  Half-life of Amlodipine
T1/2 of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Half-life of Atorvastatin
T1/2 of 2-hydroxy atorvastatin | 0 hour ~ 72 hour after drug administration
  Half-life of 2-hydroxy atorvastatin
clearance of Candesartan | 0 hour ~ 72 hour after drug administration
  Apparent clearance of Candesartan
clearance of Amlodipine | 0 hour ~ 72 hour after drug administration
  Apparent clearance of Amlodipine
clearance of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Apparent clearance of Atorvastatin
clearance of 2-hydroxy atorvastatin | 0 hour ~ 72 hour after drug administration
  Apparent clearance of 2-hydroxy atorvastatin
Vd/F of Candesartan | 0 hour ~ 72 hour after drug administration
  Apparent volume of distribution of Candesartan
Vd/F of Amlodipine | 0 hour ~ 72 hour after drug administration
  Apparent volume of distribution of Amlodipine
Vd/F of Atorvastatin | 0 hour ~ 72 hour after drug administration
  Apparent volume of distribution of Atorvastatin
Vd/F of 2-hydroxy atorvastatin | 0 hour ~ 72 hour after drug administration
  Apparent volume of distribution of 2-hydroxy atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Seunghun Han, Ph.D., Principal Investigator — Department of Clinical Pharmacology, Seoul ST.Mary's Hospital
Locations (1):
- Seoul Saint Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No